CLINICAL TRIAL: NCT00788060
Title: A Single Arm, Phase Ib Study of RAD001 and Sunitinib in Patients With Advanced Renal Cell Carcinoma
Brief Title: A Phase Ib Study of Rad001 and Sutent to Treat Renal Cell Carcinoma
Acronym: Rad/Sutent
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daniel George, MD (Other)
Collaborators: Novartis (Industry); Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Daniel George, MD, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00000548
Record Dates: First submitted 2008-11-06; First posted 2008-11-10 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma; Rad001; Sutent
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Everolimus; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RAD001 (Experimental)
  Interventions: Drug: Everolimus (RAD001); Drug: Sunitinib (Sutent)

INTERVENTIONS:
Drug: Everolimus (RAD001) — 5mg per day, continuously
  Other Names: RAD001
Drug: Sunitinib (Sutent) — 37.5 mg per day, 14 days on, 7 day break
  Other Names: Sutent

SUMMARY:
This is a single center, Phase Ib study of Sunitinib and RAD001 in patients with advanced RCC. The study design is a phase I interpatient dose-escalation with a dose expansion at the maximum tolerated dose (MTD) in patients with metastatic RCC . In the dose escalation portion, patients will be treated with sunitinib, given in an intermittent schedule (2 weeks of daily dosing followed by one week off drug. RAD001 will be given daily. Escalation of both drugs will occur as tolerated. Treatment will be arbitrarily divided into 3-week cycles, with dose limiting toxicity (DLT) determined by Cycle 2 Day 0.

DETAILED DESCRIPTION:
Escalation of both drugs will occur as tolerated. Treatment will be arbitrarily divided into 3-week cycles, with dose limiting toxicity (DLT) determined by Cycle 2 Day 0. Dose levels will be evaluated one at a time beginning with 3 patients. If 1/3 patients demonstrate DLT (as defined in section Complete), then enrollment will proceed to the next dose level. 1/3 patients develops a DLT, then 3 more patients will be accrued to this dose level. If 0-1/6 patients demonstrate DLT, then enrollment will proceed to the next dose level. However, if 2 or more patients out of 6 demonstrate DLT at a dose level, then enrollment will proceed at the next lowest dose level. The highest dose level not resulting in greater than 1/6 DLT will be considered the MTD. Dose expansion will then proceed at this dose level.

Once the maximum tolerated dose has been established for this regimen a dose expansion of 20 patients with metastatic RCC will be undertaken. Up to 10 patients with a positive FDG- PET scan at baseline (defined by 1 or more target lesions demonstrating an SUV > 5.0) will begin treatment per Figure 2B. Patients 1-10 will begin Sunitinib on Day 0 and begin RAD001 on Day 14 after repeat FDG-PET scan. Patients 11-20, will have a 2 week lead-in period of RAD001 and will begin Sunitinib 2 weeks later on Day 0. After repeat FDG-PET scan. Both groups of patients will repeat PET scan at Day 14 of cycle 2. Patients with negative FDG PET scans (SUV < 5.0 in all lesions) will not undergo repeat scanning. Patients will undergo evaluations for tumor response every 12 weeks with appropriate measurement studies (CT, MRI, bone scan). In the setting of a mixed response (progressive disease in 1 or more lesions but continued regression or stable disease below baseline in other lesions) patients may continue on study if it is determined by the PI, treating physician and patient that there is ongoing clinical benefit to the patient.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for inclusion in this study only if all of the following criteria apply:

* Patients must have histologically confirmed diagnosis of RCC.
* Patients must have undergone a nephrectomy
* Clinical or radiographic evidence of metastatic disease.
* A minimum of 4 weeks from full field radiation therapy, surgery, chemotherapy or other investigational agent. Treatment may begin one week following limited field radiation therapy.
* Subjects who have received prior limited field radiotherapy, biologic/immunotherapy or surgery must have a documented recovery period > 2 weeks
* Patients must have normal organ and marrow function as defined below:

hemoglobin > 9.0g/dL absolute neutrophil count > 1,500/μl platelets > 100,000/μl total bilirubin < 1.5 X upper limit of normal (ULN) AST(SGOT)/ALT(SGPT) < 2.5 X ULN creatinine < 1.5 X ULN (or 24 hour measured creatinine clearance > 40 mL/min) total fasting cholesterol < 350 total triglycerides < 300

* Age > 18 years.
* ECOG score of 0-2 (See Appendix 11.1).
* For patients with diabetes a Hgb A1C of ≤ 8
* Subject agrees to use a medically acceptable form of birth control during and for at least 3 months after completion of the study treatment, if he/she is sexually active
* Women of childbearing potential must have a negative serum pregnancy test within 3 days prior to treatment
* Ability to swallow and retain oral medication.
* Ability to understand and the willingness to sign a written informed consent document.
* Written informed consent obtained according to local guidelines

Exclusion Criteria:

A patient will not be eligible for inclusion in this study if any of the following criteria apply:

* History of solid organ or stem cell transplantation. Also, no current use of chronic immunosuppressive therapy is allowed.
* Patients with active brain metastases (or history of brain metastases) should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of HIV, hepatitis B, or hepatitis C infection.
* Patients who have received investigational, biologic, hormonal (other than ADT), immunotherapy, or chemotherapy less than 4 weeks prior to entry on this study or have not recovered from the toxic effects of such therapy.
* Patients who have experienced severe trauma or undergone major surgery within 4 weeks prior to entry on this study or have not recovered to grade 1 or less may not participate.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (requiring antifungal, antibiotic or antiviral therapy), symptomatic congestive heart failure (NYHC II or greater), unstable angina pectoris, cardiac arrhythmia (uncontrolled SVT or any VT), uncontrolled diabetes or psychiatric illness/social situations that would limit compliance with study requirements.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection).
* Patients who have received prior treatment with an mTOR inhibitor.
* Patients who have received prior treatment with Sunitinib are not eligible to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD)/recommended Phase 2 regimen of 2+1 dosing with Sunitinib and daily RAD001 in patients with advanced renal cell carcinoma. | 1 year
To determine the safety and tolerability of 2+1 dosing of Sunitinib and daily RAD001 in patients with advanced RCC | 1 year
To more fully evaluate the safety and tolerability of 2+1 dosing of Sunitinib and daily RAD001 at the MTD/recommended Phase 2 dose in patients with advanced RCC | 1 year

SECONDARY OUTCOMES:
Describe the non-dose limiting toxicities associated with combination therapy using 2+1 dosing Sunitinib and daily RAD001. | 1 year
Describe the pharmacokinetics of Sunitinib and RAD001 and evaluate any association with disease response | 1 year
To estimate objective response rate (partial or complete) seen in patients with advanced RCC in a dose expansion cohort treated at the MTD or recommended Phase 2 dose regimen | 1 year
To estimate the overall survival of RCC patients treated with Sunitinib and RAD001 | 1 year
To estimate the time to disease progression of RCC patients treated with Sunitinib and RAD001 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. George, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States